CLINICAL TRIAL: NCT05712174
Title: A Phase II Study of Fluorine-18 (18F)-Labeled PSMA-1007 in Patients With Known or Suspected Metastatic Prostatic Carcinoma
Brief Title: A Study of [18]F-PSMA-1007 in Patients With Known or Suspected Metastatic Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Accrual to the biochemically recurrent and metastatic cohorts complete; however, accrual to the remaining two cohorts was lagging and deemed no longer feasible.
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IIT-0030
Record Dates: First submitted 2023-01-17; First posted 2023-02-03 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Oncology; Prostate Cancer
Keywords: PSMA; [18]F-PSMA-1007; Positron Emission Tomography
MeSH Terms: conditions — Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- [18]F-PSMA-1007 PET/CT or PET/MRI (Experimental): All participants will undergo a single [18]F-PSMA-1007 PET/CT or PET/MRI scan. Intravenous bolus injection of 4 MBq/kg +/- 10% of [18]F-PSMA-1007, up to a maximum of 400 MBq.
  Interventions: Drug: [18]F-PSMA-1007

INTERVENTIONS:
Drug: [18]F-PSMA-1007 — [18]F-PSMA-1007 is a diagnostic radiopharmaceutical for use with PET/CT or PET/MRI scanning to diagnose prostate cancer.

SUMMARY:
A [18]F-PSMA-1007 PET/CT or PET/MRI scan are nuclear medicine tests used to create pictures of the whole body that may show where cells that express Prostate-Specific Membrane Antigen (PSMA) are found. PSMA is a transmembrane protein that is overexpressed in the majority of prostate cancers. PSMA imaging utilizes this overexpression, by binding on the transmembrane receptor and internalization in the cancer cells. The internalized isotope can then be imaged with the use of a PET/CT or PET/MRI scanner and show where cancer cells may be present in the body. This imaging modality has been shown to be superior to conventional imaging, such as bone scan and CT, in the detection of prostate cancer tumors.

The purpose of this study is to: 1) assess the clinical impact of a [18]F-PSMA-1007 scan on patient management plans; 2) assess the diagnostic effectiveness of a [18]F-PSMA-1007 scan in participants with known or suspected metastatic prostate cancer, as compared to standard of care CT chest, abdomen, pelvis and bone scan; 3) evaluate the safety of [18]F-PSMA-1007; and 4) assess potential correlations of PSMA level of uptake in certain tumors with cancer biologic markers such as PSA and Gleason score.

DETAILED DESCRIPTION:
This is a Phase II, diagnostic imaging, controlled, open-label, single site study in four cohorts of patients with known or suspected metastatic prostate cancer. All participants will be imaged with [18]F-PSMA-1007 PET/CT; [18]F-PSMA-1007 PET/MRI may be performed instead of a PET/CT, if PET/MRI is available.

The patients will be assessed for AEs after administration of [18]F-PSMA-1007, during their visit to the Nuclear Medicine Department. The assessment of impact on patient management will be performed using a questionnaire both before and after the [18]F-PSMA-1007 PET/CT or PET/MRI scan. The efficacy evaluation will consist of [18]F-PSMA-1007 PET/CT or PET/MRI clinical accuracy compared to standard of care CT and bone scan. Standard gadolinium-based contrast enhanced PET/MRI imaging may be performed if clinically indicated and if there are no contraindications. If a PET/MRI is performed, the clinical accuracy of the MRI component of the PET/MRI will be compared to the baseline CT. [18]F-PSMA-1007 uptake (SUVmax, Uptake Score) will be assessed in a selection of lesions and compared to PSA values collected on the day of the scan and Gleason score collected from the participant's medical history.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed prostate cancer by histopathology or cytology;
2. Eastern Cooperative Oncology Group (ECOG) Performance Scale Score ≤ 2 within two weeks of enrollment;
3. Males at least 18 years of age;
4. Any of the following clinical criteria:

   * High risk localized, treatment naive prostate cancer, defined as clinical ≥T3a, Gleason score ≥8 (or grade group 4-5), or PSA >20ng/mL. Clinical T-stage may be defined based on physical exam or standard pelvic imaging (MRI/CT).
   * High-tier intermediate risk, defined as at least two of the following: clinical T2c, Gleason score ≥7 (or Grade group 2-3) and PSA 10-20 ng/mL.
   * Biochemically recurrent prostate cancer defined as persistently elevated or rising PSA after radical prostatectomy, with a PSA value of ≥0.2ng/mL on at least two readings, or PSA with a rise of at least ≥2 ng/mL above the nadir in patients who have received definitive radiation therapy (28).
   * Metastatic disease documented on conventional imaging (CT and/or bone scan).
5. 99m-Technecium bone scan and CT of the chest abdomen and pelvis, within 4 weeks of study enrollment.
6. Receipt of a complete [18]F-PSMA-1007 PET/CT or PET/MRI referral package, including baseline history information and treatment intent from the referring physician, prior to enrolment.
7. Able and willing to follow instructions and comply with the protocol;
8. Ability to provide written informed consent prior to participation in the study.

Exclusion Criteria:

1. Inability to lie still for the entire imaging time (e.g. cough, severe arthritis, etc.);
2. Inability to complete the investigational imaging examinations due to other reasons (severe claustrophobia, radiation phobia, etc.);
3. Weight exceeding the PET/CT or PET/MRI scanner limit;
4. Known allergic reaction to [18]F-PSMA-1007;
5. Patients who have initiated new therapy (ADT, systemic therapy, or radiation) for their prostate cancer within 4 weeks of enrollment in those with high-tier intermediate risk or high risk localized prostate cancer, or biochemically recurrent prostate cancer post-prostatectomy or definitive radiotherapy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2023-09-14 (Actual); Primary Completion 2025-05-05 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
Questionnaire based assessment of the impact of [18]F-PSMA-1007 PET/CT or PET/MRI on patient management plans | Prior to and within 30 days following [18]F-PSMA-1007 PET/CT or PET/MRI
  There is sparsity of evidence regarding the impact of the results of [18]F-PSMA-1007 PET/CT or PET/MRI on patient management. With this analysis we will study whether the treatment plan is modified with the findings of the [18]F-PSMA-1007 PET/CT or PET/MRI, by asking the referring physician to complete a questionnaire on paper or electronically (via REDCap). Questions will include the patient's clinical TNM stage, treatment intent (curative vs palliative), planned treatment modalities, and clinical confidence in their treatment plan, both before and after [18]F-PSMA-1007 imaging.

SECONDARY OUTCOMES:
To confirm the diagnostic effectiveness of [18]F-PSMA-1007 PET/CT or PET/MRI in participants with known or suspected metastatic prostate cancer compared to standard of care cross-sectional imaging (CT chest, abdomen, pelvis) | Within 7 days post [18]F-PSMA-1007 PET/CT or PET/MRI
  A Nuclear Medicine physician will correlate the [18]F-PSMA-1007 PET/CT or PET/MRI findings with CT findings and comment on whether [18]F-PSMA-1007 avid lesions are visualized on standard of care imaging. The [18]F-PSMA-1007 PET/CT or PET/MRI scan findings will be compared globally to standard of care imaging to document if more or fewer lesions are seen on [18]F-PSMA-1007 PET/CT or PET/MRI than conventional imaging.
  A reader confidence score will be used to assess reader certainty in finding characterization. The findings will be considered metastatic for scores 4 and 5.
To confirm the diagnostic effectiveness of [18]F-PSMA-1007 PET/CT or PET/MRI in participants with known or suspected metastatic prostate cancer compared to standard of care cross-sectional imaging (bone scan) | Within 7 days post [18]F-PSMA-1007 PET/CT or PET/MRI
  A Nuclear Medicine physician will correlate the [18]F-PSMA-1007 PET/CT or PET/MRI findings with bone scan findings and comment on whether [18]F-PSMA-1007 avid lesions are visualized on standard of care imaging. The [18]F-PSMA-1007 PET/CT or PET/MRI scan findings will be compared globally to standard of care imaging to document if more or fewer lesions are seen on [18]F-PSMA-1007 PET/CT or PET/MRI than conventional imaging.
  A reader confidence score will be used to assess reader certainty in finding characterization. The findings will be considered metastatic for scores 4 and 5.
The [18]F-PSMA-1007 level of avidity will be assessed in selected lesions and compared to background activity and cancer biologic markers (PSA value) | Within 7 days post [18]F-PSMA-1007 PET/CT or PET/MRI
  We will explore whether there is a correlation between [18]F-PSMA-1007 uptake and PSA values. The intensity of tumor uptake of [18]F-PSMA-1007 will be assessed by an experienced Nuclear Medicine physician using visual interpretation and computer-assisted techniques in up to five (5) lesions. The maximum Standardized Uptake Value (SUVmax) will be determined for the tumor site(s), the liver, blood pool and parotid using the standard algorithm available on the PET scanners.
The [18]F-PSMA-1007 level of avidity will be assessed in selected lesions and compared to background activity and cancer biologic markers (Gleason score) | Within 7 days post [18]F-PSMA-1007 PET/CT or PET/MRI
  We will explore whether there is a correlation between [18]F-PSMA-1007 uptake and Gleason score. The intensity of tumor uptake of [18]F-PSMA-1007 will be assessed by an experienced Nuclear Medicine physician using visual interpretation and computer-assisted techniques in up to five (5) lesions. The maximum Standardized Uptake Value (SUVmax) will be determined for the tumor site(s), the liver, blood pool and parotid using the standard algorithm available on the PET scanners.
To evaluate the safety of [18]F-PSMA-1007 PET/CT or PET/MRI imaging | Up to 24 hours after [18]F-PSMA-1007 administration
  Adverse events (AEs) following [18]F-PSMA-1007 administration will be assessed and graded using CTCAE v.5.

CONTACTS AND LOCATIONS:
Overall Officials: Stella Koumna, MD, Principal Investigator — Cross Cancer Institute, Alberta Health Services
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No